CLINICAL TRIAL: NCT02370563
Title: An Open-Label Study of the Efficacy of 18F-FSPG PET/CT in Subjects With Intracranial Cancers
Brief Title: PET Imaging of Intracranial Cancers With 18F-FSPG
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Life Molecular Imaging SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FSPG010114
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Brain Cancer
MeSH Terms: conditions — Brain Neoplasms | interventions — 4-(3-fluoropropyl)glutamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): 18F-FSPG will be administered to 30 patients with brain tumors or brain metastases.
  Interventions: Drug: 18F-FSPG

INTERVENTIONS:
Drug: 18F-FSPG — 18F-FSPG is a novel F18-labelled, radiopharmaceutical agent for PET imaging. It is administered intravenously at a dose of 300 MBq (8.1mCi ± 10%).

SUMMARY:
The aim of this study is to explore the efficacy of 18F-FSPG in the detection of primary or metastatic brain cancer lesions confirmed by a standard of truth, preferably histology. This is a single center, open labelled, non-randomized study. A total of 30 subjects with brain tumor or brain metastases will be enrolled. All different stages of malignancies will be recruited, including those with different types of pathologies and grades, and newly diagnosed or recurrent disease.

DETAILED DESCRIPTION:
Subjects with various types and grades of primary brain tumors or brain metastasis will be recruited. The brain tumor needs to be either histologically or clinically confirmed. 18F-FSPG will be injected intravenously into the subjects, and PET/CT imaging performed. Images will be assessed visually and quantitatively.

Available tumor specimens will be analyzed by immunohistochemistry (IHC) for example for expression of components of the system xc- and associated biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Participant must be able to complete a PET/CT scan and MRI without the use of sedation
3. Participant has

   * a primary brain tumor that has been histologically confirmed
   * OR confirmed or suspected recurrent brain cancer or brain metastasis for which the primary tumor has been histologically confirmed,
   * OR a brain lesion that is concerning for malignancy for which histopathological confirmation is anticipated following enrollment (e.g., biopsy or surgical resection of the tumor is scheduled)
   * OR a suspected low-grade brain tumor, where confirmation is based upon a combination of other imaging (e.g. PET/CT, MRI, diagnostic CT) and clinical assessment.
   * All pathology specimens must be within 1 year of the planned 18F-FSPG PET/CT scan.
4. The time interval between 18F-FSPG PET/CT and other imaging (including other PET/CTs, MRI or diagnostic CT) should be within 4 weeks (exceptions will be allowed for 6 weeks, if there are no other options)
5. Karnofsky Performance Status Scale of 60 or higher OR an ECOG Performance Status of 0-2.
6. No clinically relevant deviations in renal function (Serum Creatinine > Grade 2 CTCAE v4.0.). Maximal interval between confirmation and injection of 18F-FSPG is one week.
7. No chemotherapy, radiotherapy, or immune/biologic therapy scheduled or performed between other imaging (PET/CTs, MRI, or diagnostic CTs) and18F-FSPG PET/CT.

Exclusion Criteria:

1. Patient is scheduled for brain surgery and/or another invasive procedure within the time period of one month prior to 18F-FSPG administration. Minimally invasive needle biopsies are allowed.
2. Known hypersensitivity to the study drug or components of the preparation
3. Patient has completed participation in another clinical study involving administration of an investigational agent in the preceding 4 weeks. However, participation in clinical studies involving other investigational PET or SPECT tracers will not be excluded if in the opinion of the Investigator:

   * evaluation of 18F-FSPG safety and tolerability will not be confounded by the other investigational PET or SPECT tracer
   * a minimum of two days (or longer as necessary based on radiological half-life) have elapsed between investigational PET or SPECT tracer administrations to allow acceptable clearance of the tracer
   * the investigational PET or SPECT tracer administration was well tolerated by the patient.
4. Investigator precludes participation for scientific reasons, for reasons of compliance (e.g., concurrent disease which could compromise the subject's study completion), or for reasons of the patient's safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Location and number of lesions and their location as detected by 18F-FSPG uptake above background in the brain of each study subject following visual inspection of the 18F-FSPG PET/CT scans | 0-75 min

SECONDARY OUTCOMES:
Location and number of lesions detected in the whole body following visual inspection of the 18F-FSPG PET/CT scans | 0-75 min
Location and number of lesions detected in the brain and whole body following visual inspection of the CT, MR or other available PET (e.g. 18F-FDG, 18F-FLT, etc.). | <4 weeks from FSPG PET/CT scan
Lesion size measured by means of ROIs drawn on (contrast-enhanced) MR or CT. | <4 weeks from FSPG PET/CT scan
18F-FSPG standardized uptake value (SUV) measured in each detected lesion and in the background (region without lesion). | 0-75 min
SUV measured in each detected lesion and in the background using other available PET tracers (e.g. 18F-FDG, 18F-FLT, etc.). | < 4 weeks from FSPG PET/CT scan
Determination of FSPG PET/CT image quality based on visual inspection. | 0-75 min

CONTACTS AND LOCATIONS:
Overall Officials: Norman Koglin, PhD, Study Director — Life Molecular Imaging SA
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

REFERENCES:
- [Derived] Wardak M, Sonni I, Fan AP, Minamimoto R, Jamali M, Hatami N, Zaharchuk G, Fischbein N, Nagpal S, Li G, Koglin N, Berndt M, Bullich S, Stephens AW, Dinkelborg LM, Abel T, Manning HC, Rosenberg J, Chin FT, Gambhir SS, Mittra ES. 18F-FSPG PET/CT Imaging of System xC- Transporter Activity in Patients with Primary and Metastatic Brain Tumors. Radiology. 2022 Jun;303(3):620-631. doi: 10.1148/radiol.203296. Epub 2022 Feb 22. PMID 35191738